CLINICAL TRIAL: NCT06863298
Title: Listen and Learn: The Effect of Podcast Use on Nursing Students' Stoma Bag Changing Knowledge and Skills: A Randomized Controlled Trial
Brief Title: Use of Podcast in Nursing Students' Stoma Bag Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Assistant Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Use of Podcasts in Nursing
Record Dates: First submitted 2025-02-27; First posted 2025-03-07 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Nurse's Role

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled trial in parallel groups. Students will be randomly divided into two groups (Control and intervention). Students in the control group will not receive any intervention other than routine education. Students in the intervention group will receive podcasting outside of routine education.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Students will know that they are in the control or intervention group. Because an agreement will be signed with the students in the intervention group that the podcast will not be shared. Since researchers other than those who signed the agreement will be doing the application, the researchers will not know which group the students are in. Since statistical blinding will also be done, the result evaluator will not know the groups of the students.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The students in the control group will first receive theoretical training on stoma and bag change. After the training, the students will be given the "Stoma Bag Change Knowledge Test". Then, the students will be given a laboratory demonstration on stoma and bag change. After this routine training, no intervention will be made in the control group. Approximately two weeks later, the students will be given a skill assessment according to the "Stoma Bag Change Skill Checklist". One week after the skill assessment, the students will be given the "Stoma Bag Change Knowledge Test" again.
- Podcast group (Experimental): The students in the intervention group will first receive theoretical training on stoma and bag change. After the training, the students will be given the "Stoma Bag Change Knowledge Test". Then, the students will be given a laboratory demonstration on stoma and bag change. After this routine training, the Podcast (about stoma and bag change) prepared by the researchers will be made available to the students in the intervention group. Students will listen to the Podcast, which will be prepared for two weeks, as many times as they want, whenever and wherever they want. After two weeks, the Podcast access will be closed and the students will be given a skill assessment according to the "Stoma Bag Change Skill Checklist". One week after the skill assessment, the "Stoma Bag Change Knowledge Test" will be applied to the students again. Finally, a "Satisfaction with the Teaching Method Survey" will be applied to determine the students' experiences regarding learning the Podcast.
  Interventions: Other: Podcast

INTERVENTIONS:
Other: Podcast — A podcast is content that can be listened to on any digital audio listening device, including a computer, that supports audio file playback.
  Arms: Podcast group

SUMMARY:
The research will be conducted to determine the effect of podcast use on nursing students' knowledge and skills on stoma bag changing. The universe of a randomized controlled study with a pre-test-post-test control group will consist of 165 first-year students enrolled in Necmettin Erbakan University Faculty of Nursing in the 2024-2025 Fall Semester. The research is planned to be completed with a total of n=80 first-year students, n=40 in the control group and n=40 in the intervention group. The selected 80 students will be randomly assigned to two groups (A and B) so that the general academic success scores of both groups will be homogeneous. The data of the research will be collected with the "Personal Information Form", "Stoma Bag Changing Knowledge Test", "Stoma Bag Changing Skills Checklist" and "Satisfaction with Teaching Method Survey". After the theoretical training on stoma, a laboratory demonstration will be given. Then, no intervention will be applied to the control group. The intervention group will listen to the Podcast prepared by the researchers. The data obtained from the research will be analyzed with the licensed SPSS 22.0 package program. It is thought that the information obtained from the research will contribute to the literature.

DETAILED DESCRIPTION:
Stoma is a common procedure used in the surgical treatment of cancers related to the gastrointestinal or urinary system, inflammatory bowel diseases and traumas. Stoma opening increases the survival rates of individuals, but stoma-related complications are considered as negative consequences of living with an ostomy. Negative effects on stoma patients are physical, psychological and social. Physical problems of stoma patients include leakage, skin problems and odor. The most common physical problems related to stoma include leakage, peristomal skin problems and the need for adaptation of stoma devices and the need to adapt clothing to the presence and location of the stoma, which has a significant impact on the patient's daily life. Stoma patient care is included in the curriculum of pre-licensure nursing programs, but the number of studies examining student nurses' knowledge of stoma care is limited. In a study, it was concluded that nursing students had initial knowledge about ostomy care and very limited clinical experience, but they were highly confident in providing ostomy care. Therefore, it is very important to develop the knowledge and skill levels of undergraduate nursing students about stoma and bag change, which plays an important role in the care of stoma patients.

In nursing education, there has been a transition from traditional pedagogical models to current methods that use technology for information acquisition. One of the teaching methodologies used in nursing education is Podcast. Podcast emerged as a result of discussions aimed at understanding and learning by listening. The term "podcast" has been in use since approximately 2004. It was originally derived from two terms, "iPod" and "broadcast." A podcast can be listened to on any digital audio listening device, including a computer that supports audio file playback. Therefore, podcasts can be listened to 24/7 and on the go. These combined qualities have significantly increased podcast use over the last 20 years. Over time, podcasts have begun to be used as an effective medical education tool. In a study, it was determined that podcasts did not affect the knowledge level of nursing students, but students were satisfied with this learning experience. Studies determining the effectiveness of podcasts on nursing students are quite limited. Studies conducted have mostly investigated the effect of podcasts on students' knowledge level and satisfaction. This study aimed to determine the effect of podcast use on nursing students' knowledge and skills regarding stoma bag change. There is no study in the literature examining the effect of podcast use on nursing students' knowledge and skills in changing stoma bags. Therefore, the research is original in its field. It is thought that the study will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Must be registered in the first year of the Faculty of Nursing,
* Must be taking the Fundamentals of Nursing course for the first time,
* Must be willing to participate in the research.

Exclusion Criteria:

* Coming through horizontal or vertical transfer,
* Having difficulty understanding and speaking Turkish,
* Being a Health Vocational High School graduate,
* Not attending theoretical training on stoma care,
* Not attending any of the research steps (Pre-test, Podcast application, post-test),
* Wanting to leave the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Stoma Bag Change Knowledge Test | Up to 1-2 months
  It was prepared by researchers in line with the theoretical course content and learning objectives regarding changing the stoma bag in line with the literature. The knowledge test consists of 20 closed-ended questions with five options that determine the knowledge level of students regarding changing the stoma bag. The distribution of the questions in the knowledge test was made according to the target behaviors of the subject. The evaluation of the knowledge test will be made out of 100 points. The knowledge test results will be evaluated as "5" points for each correct answer and "0" points for each wrong answer. In this context, the lowest score that students can get from the knowledge test will be "0" and the highest score will be "100" points.
Stoma Bag Changing Skills Checklist | up to 2 months
  In order to evaluate the students' skills in changing the stoma bag (determination of the materials to be used and correct implementation of the application), it was prepared by researchers in line with the literature. The skill checklist consists of 25 steps. Each step is aimed at evaluating the application as correct/complete, incorrect/incomplete and not implemented. The skill checklist was prepared in line with the stoma bag changing skill guide used in the laboratory demonstration application of the students. In the skill checklist, if the skill application was performed correctly/completely, it will be evaluated as 2 points, if it was incorrect/incomplete/completed, it will be evaluated as "1" point and if it was not implemented, it will be evaluated as "0" point. In this context, students can get the lowest "0" point and the highest "50" point from the skill checklist.
Satisfaction Survey on Teaching Methods | up to 2 months
  It consists of seven questions on a 5-point Likert scale prepared by the researchers in line with the literature in order to evaluate the satisfaction of the students in the intervention group regarding learning through the use of Podcast.

CONTACTS AND LOCATIONS:
Locations (1):
- Neu University, Konya, Turkey (Türkiye)